CLINICAL TRIAL: NCT01204879
Title: Reinforcing Exercise in Substance Abusing Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-010S-2; R01DA027615 (NIH)
Record Dates: First submitted 2010-08-09; First posted 2010-09-17 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2016-12

CONDITIONS: Substance Abuse; Contingency Management; Exercise
MeSH Terms: conditions — Substance-Related Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CM for general activities (Active Comparator): Standard care plus individual contingency management session for general activities
  Interventions: Behavioral: Contingency Management
- CM for exercise-related activities (Experimental): Standard care plus individual contingency management session for physical activities
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Participants earn the chance to win prizes for the targeted behavior.

SUMMARY:
This study will evaluate the efficacy of an exercise-based contingency management (CM) intervention. A total of 120 substance abusing patients in intensive outpatient treatment will be randomly assigned to one of two conditions: (a) standard care plus CM for completing goal-related activities not related to exercising (e.g., improving work, family, or transportation issues), or (b) standard care plus CM for completing exercise-related activities. Compared to those receiving goal-related CM activity contracting, it is expected that those in the exercise CM condition will participate in more physical activities and develop greater strength and flexibility, decrease drug use, reduce HIV risk behaviors, lessen depressive symptoms, and improve health indices.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years
* English speaking
* in substance abuse treatment
* written permission from a physician (or their designated health care professional, e.g., nurse, physicians assistant) to participate in the study and an exercise program.

Exclusion Criteria:

* inability to comprehend the study
* in recovery for pathological gambling
* contraindication for exercising

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
physical activity participation and functioning measured by the PAQ (Kcal/wk expenditures) | baseline
physical activity participation and functioning measured by the PAQ (Kcal/wk expenditures) | month 2
physical activity participation and functioning measured by the PAQ (Kcal/wk expenditures) | month 4
physical activity participation and functioning measured by the PAQ (Kcal/wk expenditures) | month 6
physical activity participation and functioning measured by the PAQ (Kcal/wk expenditures) | month 9
physical activity participation and functioning measured by the PAQ (Kcal/wk expenditures) | month 12
attendance at exercise classes | baseline
attendance at exercise classes | month 2
attendance at exercise classes | month 4
attendance at exercise classes | month 6
attendance at exercise classes | month 9
attendance at exercise classes | month 12

SECONDARY OUTCOMES:
longest duration of abstinence | baseline
longest duration of abstinence | month 2
longest duration of abstinence | month 4
longest duration of abstinence | month 6
longest duration of abstinence | month 9
longest duration of abstinence | month 12
HIV risk behaviors as reported on HRBS questionnaire | baseline
HIV risk behaviors as reported on HRBS questionnaire | month 2
HIV risk behaviors as reported on HRBS questionnaire | month 4
HIV risk behaviors as reported on HRBS questionnaire | month 6
HIV risk behaviors as reported on HRBS questionnaire | month 9
HIV risk behaviors as reported on HRBS questionnaire | month 12
psychological distress as reported on BSI questionnaire | baseline
psychological distress as reported on BSI questionnaire | month 2
psychological distress as reported on BSI questionnaire | month 4
psychological distress as reported on BSI questionnaire | month 6
psychological distress as reported on BSI questionnaire | month 9
psychological distress as reported on BSI questionnaire | month 12

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — University of Conncecticut Health Center
Locations (1):
- Alcohol and Drug Recovery Centers, Inc., Hartford, Connecticut, United States